CLINICAL TRIAL: NCT04138472
Title: Comparison Of Dexmedetomidine, Fentanyl And Lignocaine In Attenuation Of Hemodynamic Response To Direct Laryngoscopy And Intubation In Patient Undergoing Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sana Urooj (Other)
Collaborators: Dow University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Sana Urooj, SUrooj, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Dexmedetomidine; Fentanyl; Lignocaine; Laryngoscopy; Hemodynamic Response; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Masking Description: Patients do not know about the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): Group A patients receive intravenous dexmedetomidine 0.06mg/kg in 100ml normal saline 0.9% over 10minutes.
  Interventions: Drug: dexmedetomidine
- Fentanyl (Experimental): Group B receives intravenous fentanyl at 2mcg/kg in 100ml saline over 10 minutes in induction room.
  Interventions: Drug: fentanyl
- Lidocaine (Experimental): Group C patients receives intravenous lidocaine 1.5mg/kg in 100ml saline over 10 minutes in induction room.
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: dexmedetomidine — intravenous dexmedetomidine 0.06mg/kg in 100ml normal saline 0.9% over 10minutes.
  Arms: Dexmedetomidine
Drug: fentanyl — intravenous fentanyl at 2mcg/kg in 100ml saline over 10 minutes in induction room.
  Arms: Fentanyl
Drug: lidocaine — intravenous lidocaine 1.5mg/kg in 100ml saline over 10 minutes in induction room.
  Arms: Lidocaine

SUMMARY:
Comparison Of Dexmedetomidine, Fentanyl And Lignocaine In Attenuation Of Hemodynamic Response To Direct Laryngoscopy And Intubation In Patient Undergoing Laparoscopic Cholecystectomy

DETAILED DESCRIPTION:
Direct laryngoscopy and intubation are painful stimulus that activates sympathoadrenal discharge which results in intense cardiovascular reflex i.e. tachycardia and hypertension. In this study we will compare effects of intravenous dexmedetomidine, fentanyl and lidocaine for attenuation of these reflexes in patient undergoing laproscopic cholecystectomy. how these agents will effect hemodynamic response during pneumoperitoneum. Tertiary objective will be to observe sedation, perioperative complications and recovery in these patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA-I and ll patients
* Male and female patient of age 20-70 years.
* Undergoing Elective surgery
* Intubation by skilled anesthetist of at least 2 years' experience
* Intubation not more than 45 seconds

Exclusion Criteria:

* Patients with uncontrolled DM, HTN, IHD, endocrine or autonomic dysfunction
* Pregnant and lactating females
* Short thick neck with anticipated difficult intubation
* Any sort of obstructive restrictive or reactive airway disease
* Patient allergic to any of the study medications.
* Obese patients, Narcotic addicts

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure | at induction
  hermodynamic response (Top number will be assessed of blood pressure)
Diastolic blood pressure | at induction
  hermodynamic response (bottom number will be assessed of blood pressure)
mean atrial pressure | at induction
  Hemodynamic responses (average blood pressure in an individual during a single cardiac cycle)
Heart rate | at induction
  Hemodynamic responses (average heart rate beats a minute)
Oxygen saturation (SpO2) | at induction
  Hemodynamic responses) (arterial oxy-hemoglobin saturation is measured non-invasively by a finger pulse oximeter or handheld pulse oximeter,

SECONDARY OUTCOMES:
Sedation assessment | at 10 minutes post operative
  Ramsey score use for sedation, it consist of 1-6 where 6 indicates worst(no response) and 6 indicates good response
Recovery assessment | at 10 minutes post operatively
  Aldret score use for recovery assessment, it consist of 0-10 point where 0 indicates worst(no response) and 10 indicates good response
Complications | 1 week Post-operative(Operation -discharge)
  Cough, Laryngospasm, Bradycardia, Regugitation, PONV, Hypertention, Hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- DUHS, Civil hospital Karachi (CHK), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No